CLINICAL TRIAL: NCT01944072
Title: Pulmonary Rehabilitation in COPD: Effects of Two Aerobic Exercise Intensity in Patient-centered Outcomes - a Randomized Controlled Trial
Brief Title: Pulmonary Rehabilitation in COPD: Effects of Two Aerobic Exercise Intensity in Patient-centered Outcomes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Nova de Lisboa (Other)
Collaborators: Centro Hospitalar Lisboa Norte (Other); Centro de Estudos de Doenças Crónicas (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: NOVA-FCM-MSAR-001
Record Dates: First submitted 2013-09-09; First posted 2013-09-17 (Estimated); Last update posted 2013-09-17 (Estimated); Status verified 2013-09

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Chronic Obstructive Pulmonary Disease; COPD; Pulmonary rehabilitation; Aerobic exercise; CEDOC; FCM; UNL; NOVA MEDICAL SCHOOL
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- 60% (Other): aerobic exercise training intensity of 60%Wmax
  Interventions: Other: Aerobic exercise training intensity
- 80% (Other): aerobic exercise training intensity of 80%Wmax
  Interventions: Other: Aerobic exercise training intensity

INTERVENTIONS:
Other: Aerobic exercise training intensity

SUMMARY:
Trial design: An equivalence/non-inferiority randomized controlled trial with parallel group design studied the effect of two aerobic exercise-training intensities in COPD patient-centered outcomes. Methods: Thirty-four COPD clinically stable patients stratified from mild to very severe GOLD stages, were blinded to 60 or 80%Wmax aerobic exercise training intensity in an outpatient pulmonary rehabilitation program, between 2009-2010. Outcomes were assessed with St.George's respiratory questionnaire (primary outcome), Mahler dyspnea index, London Chest activity of daily living scale, 6-minute walk, constant load and incremental exercise tests. Patient's allocation sequence was computer-generated, with consignment in a safe deposit box.

ELIGIBILITY:
Inclusion Criteria:

* Clinically stable COPD
* FEV1/FVC < 70%
* Exercise training medical referral

Exclusion Criteria:

* Unable to attend 3-times/week program
* Infectious disease
* Metastatic cancer
* Unstable heart disease
* Neuromusculoskeletal disorder
* Cognitive or psychiatric disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2009-09; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Health-related quality-of-life measured by the St.George's respiratory questionnaire | 8 weeks (20 sessions)

SECONDARY OUTCOMES:
Symptoms control measured by the Mahler dyspnea index | 8 weeks (20 sessions)
Exercise Tolerance | 8 weeks (20 sessions)
  exercise tolerance assessed by the London-Chest activity of daily-living scale, 6-minute walk test, incremental exercise test and constant-load exercise test

CONTACTS AND LOCATIONS:
Overall Officials: Catarina Santos, PT, MSc, Principal Investigator — Centro Hospitalar Lisboa Ocidental; Fátima Rodrigues, MD, MSc, Study Chair — Centro Hospitalar Lisboa Norte; Cristina Bárbara, MD, PhD, Study Director — Centro Hospitalar Lisboa Norte

REFERENCES:
- [Derived] Santos C, Rodrigues F, Santos J, Morais L, Barbara C. Pulmonary Rehabilitation in COPD: Effect of 2 Aerobic Exercise Intensities on Subject-Centered Outcomes--A Randomized Controlled Trial. Respir Care. 2015 Nov;60(11):1603-9. doi: 10.4187/respcare.03663. Epub 2015 Jul 28. PMID 26221044